CLINICAL TRIAL: NCT01161472
Title: A 4 Way Placebo And Active Controlled Study To Evaluate The Effects Of Fesoterodine On Cognitive Function In Healthy Elderly Subjects
Brief Title: A Study to Assess the Cognitive Effects of Fesoterodine in Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: A0221086
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
MeSH Terms: interventions — fesoterodine; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 4mg fesoterodine (Experimental)
  Interventions: Drug: 4mg fesoterodine
- fesoterodine 8mg (Experimental)
  Interventions: Drug: 8mg fesoterodine
- 1mg alprazolam (Active Comparator)
  Interventions: Drug: alprazolam 1mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4mg fesoterodine — 4mg tablet once daily for 6 days
  Arms: 4mg fesoterodine
Drug: 8mg fesoterodine — 4mg tablet once daily for 3 days followed by 8mg tablet once daily for 3 days
  Arms: fesoterodine 8mg
Drug: alprazolam 1mg — 1mg tablet once on last day of treatment period at clinic
  Arms: 1mg alprazolam
Drug: Placebo — Placebo tablet for fesoterodine once daily for 6 days and placebo tablet for alprazolam once on last day of treatment period at clinic
  Arms: Placebo

SUMMARY:
The study is designed to evaluate elements of cognitive function in subjects receiving either fesoterodine or alprazolam.

DETAILED DESCRIPTION:
Evaluation of cognitive function

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers 65 years and over with minimum MMSE of 26

Exclusion Criteria:

* Prohibited concomitant medications
* Confounding medical conditions
* Clinically significant comorbid diseases
* Hypersensitivity or contraindications to fesoterodine or active control

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221086&StudyName=A%20study%20to%20assess%20the%20cognitive%20effects%20of%20fesoterodine%20in%20elderly%20subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg: Fesoterodine 4 milligram (mg) tablet administered orally once daily (OD) for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the first intervention period; followed by placebo matched to fesoterodine 4 mg or 8 mg tablet orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the second intervention period; then fesoterodine 4 mg tablet administered orally OD for the first 3 days followed by fesoterodine 8 mg tablet orally OD for the next 3 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the third intervention period; and placebo matched to fesoterodine 4 mg or 8 mg tablet administered orally OD for 6 days along with a single oral dose of alprazolam 1 mg capsule on Day 6 in the fourth intervention period. A washout period of at least 3 to 6 days was maintained between each treatment period.
- Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo: Fesoterodine 4 mg tablet administered orally OD for the first 3 days followed by fesoterodine 8 mg tablet orally OD for the next 3 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the first intervention period; then fesoterodine 4 mg tablet administered orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the second intervention period; followed by placebo matched to fesoterodine 4 mg or 8 mg tablet administered orally OD for 6 days along with a single oral dose of alprazolam 1 mg capsule on Day 6 in the third intervention period; and placebo matched to fesoterodine 4 mg or 8 mg tablet orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the fourth intervention period. A washout period of at least 3 to 6 days was maintained between each treatment period.
- Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg: Placebo matched to fesoterodine 4 mg or 8 mg tablet administered orally OD for 6 days along with a single oral dose of alprazolam 1 mg capsule on Day 6 in the first intervention period; followed by fesoterodine 4 mg tablet administered orally OD for the first 3 days followed by fesoterodine 8 mg tablet orally OD for the next 3 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the second intervention period; then placebo matched to fesoterodine 4 mg or 8 mg tablet orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the third intervention period; and fesoterodine 4 mg tablet administered orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the fourth intervention period. A washout period of at least 3 to 6 days was maintained between each treatment period.
- Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg: Placebo matched to fesoterodine 4 mg or 8 mg tablet orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the first intervention period; followed by placebo matched to fesoterodine 4 mg or 8 mg tablet administered orally OD for 6 days along with a single oral dose of alprazolam 1 mg capsule on Day 6 in the second intervention period; then fesoterodine 4 mg tablet administered orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the third intervention period; and fesoterodine 4 mg tablet administered orally OD for the first 3 days followed by fesoterodine 8 mg tablet orally OD for the next 3 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in the fourth intervention period. A washout period of at least 3 to 6 days was maintained between each treatment period.
Period: First Intervention Period
Arm/Group | Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg | Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo | Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg | Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg
Started | 5 | 5 | 5 | 5
Treated | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (At Least 3 to 6 Days)
Arm/Group | Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg | Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo | Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg | Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg | Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo | Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg | Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (At Least 3 to 6 Days)
Arm/Group | Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg | Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo | Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg | Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg
Started | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg | Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo | Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg | Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (At Least 3 to 6 Days)
Arm/Group | Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg | Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo | Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg | Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | Fesoterodine 4 mg, Placebo, Fesoterodine 8 mg, Aplrazolam 1 mg | Fesoterodine 8 mg, Fesoterodine 4 mg, Aplrazolam 1 mg, Placebo | Aplrazolam 1 mg, Fesoterodine 8 mg, Placebo, Fesoterodine 4 mg | Placebo, Aplrazolam 1 mg, Fesoterodine 4 mg, Fesoterodine 8 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All participants randomized to any treatment (fesoterodine 4 mg tablet first, fesoterodine 8 mg tablet first, alprazolam 1 mg capsule first and placebo first).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Computer Based Objective Cognition Testing (CogState) Detection Speed
Description: Detection speed: a cognitive test which assessed psychomotor function. A playing card was presented face up in the center of the screen. As soon as this happened, the participant was to press the 'Yes' key. The outcome measure was speed of performance; mean of the log10 transformed reaction time for correct responses [measured in log10 milliseconds (MS)]. Lower scores meant a better performance.
Time Frame: Baseline
Population: The Per Protocol (PP) Analysis Set included all randomized participants who completed the study, received treatment in all 4 study periods until the end of treatment visit in the fourth study period and who were not serious protocol violators. 'N' (Number of participants analyzed) signifies participants evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: Log10 MS
Groups:
- Fesoterodine 4 mg: Fesoterodine 4 mg tablet administered orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in any of the intervention periods.
- Fesoterodine 8 mg: Fesoterodine 4 mg tablet administered orally OD for the first 3 days followed by fesoterodine 8 mg tablet orally OD for the next 3 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in any of the intervention periods.
- Aplrazolam 1 mg: Placebo matched to fesoterodine 4 mg or 8 mg tablet administered orally OD for 6 days along with a single oral dose of alprazolam 1 mg capsule on Day 6 in any of the intervention periods.
- Placebo: Placebo matched to fesoterodine 4 mg or 8 mg tablet orally OD for 6 days along with placebo matched to a single oral dose of alprazolam 1 mg capsule on Day 6 in any of the intervention periods.
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Log10 MS | 2.6333 (0.1049) | 2.5971 (0.0937) | 2.6103 (0.1107) | 2.5842 (0.0875)

2. Primary Outcome: Change From Baseline in Computer Based Objective Cognition Testing (CogState) Detection Speed on Day 6
Description: as for outcome 1
Time Frame: Baseline and Day 6
Population: The PP Analysis Set included all randomized participants who completed the study, received treatment in all 4 study periods until the end of treatment visit in the fourth study period and who were not serious protocol violators. 'N' (Number of participants analyzed) signifies participants evaluable for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Log10 MS
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Log10 MS | -0.0201 (0.0153) | -0.0119 (0.0150) | 0.0684 (0.0150) | 0.0084 (0.0152)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg vs Placebo; Analysis of Covariance (ANCOVA) was used to determine p-value for comparison of fesoterodine 4 mg vs placebo, with model terms: period and treatment as the fixed effect, participants as the random effect, and between and within participant baselines as the covariates; Test type: Superiority or Other; p = 0.1198, ANCOVA; Least square (LS) Mean Difference = -0.0285, 95% CI 2-sided [-0.0647 to 0.0077], Standard Error of Mean 0.0180
Statistical Analysis 2: Comparison: Fesoterodine 8 mg vs Placebo; ANCOVA was used to determine p-value for comparison of fesoterodine 8 mg vs placebo, with model terms: period and treatment as the fixed effect, participants as the random effect, and between and within participant baselines as the covariates; Test type: Superiority or Other; p = 0.2459, ANCOVA; LS Mean Difference = -0.0203, 95% CI 2-sided [-0.0551 to 0.0145], Standard Error of Mean 0.0173

3. Secondary Outcome: CogState Identification Speed
Description: Identification speed: a cognitive test which assessed visual attention. A playing card was presented face up in the center of the screen. As soon as this happened, the participant had to decide whether the card was red or not. The outcome measure was speed of performance; mean of the log10 transformed reaction time for correct responses (measured in log10 MS). Lower scores meant a better performance.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 MS
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Log10 MS | 2.7540 (0.0505) | 2.7672 (0.0610) | 2.7577 (0.0577) | 2.7457 (0.0637)

4. Secondary Outcome: Change From Baseline in CogState Identification Speed on Day 6
Description: as for outcome 3
Time Frame: Baseline and Day 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Log10 MS
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Log10 MS | 0.0105 (0.0084) | 0.0057 (0.0085) | 0.0817 (0.0084) | 0.0142 (0.0085)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg vs Placebo; ANCOVA was used to determine p-value for comparison of fesoterodine 4 mg vs placebo, with model terms: period and treatment as the fixed effect, participants as the random effect, and between and within participant baselines as the covariates; Test type: Superiority or Other; p = 0.7502, ANCOVA; LS Mean Difference = -0.0037, 95% CI 2-sided [-0.0268 to 0.0194], Standard Error of Mean 0.0115
Statistical Analysis 2: Comparison: Fesoterodine 8 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4785, ANCOVA; LS Mean Difference = -0.0085, 95% CI 2-sided [-0.0325 to 0.0154], Standard Error of Mean 0.0119

5. Secondary Outcome: CogState One Card Learning
Description: One card learning: a cognitive test which assessed visual learning. Participants were to remember which cards were previously shown in a task. The outcome measure was accuracy of performance; arcsine transformation of the square root (sqrt) of the proportion of correct responses. Higher scores meant a better performance.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Arcsine [(sqrt) proportion correct]
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Arcsine [(sqrt) proportion correct] | 0.9585 (0.0893) | 0.9421 (0.0878) | 0.9531 (0.1062) | 0.9302 (0.0822)

6. Secondary Outcome: Change From Baseline in CogState One Card Learning on Day 6
Description: as for outcome 5
Time Frame: Baseline and Day 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Arcsine [(sqrt) proportion correct]
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Arcsine [(sqrt) proportion correct] | -0.0094 (0.0204) | 0.0151 (0.0203) | -0.0880 (0.0204) | -0.0058 (0.0205)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.8944, ANCOVA; LS Mean Difference = -0.0035, 95% CI 2-sided [-0.0569 to 0.0498], Standard Error of Mean 0.0265
Statistical Analysis 2: Comparison: Fesoterodine 8 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4308, ANCOVA; LS Mean Difference = 0.0209, 95% CI 2-sided [-0.0320 to 0.0738], Standard Error of Mean 0.0263

7. Secondary Outcome: CogState Continuous Paired Associate Learning (CPAL)
Description: CPAL: a cognitive test which assessed visual episodic learning. Participant was to learn and remember picture locations on the screen and was to tap the target on the central location to begin. As each picture was revealed, the participant was to remember where the picture was located and tap that location. The outcome measure was the number of errors made in correctly placing each of the 4 patterns in their location 4 times. Lower scores meant a better performance.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Errors | 96.33 (57.058) | 99.83 (55.343) | 89.50 (58.240) | 107.44 (53.388)

8. Secondary Outcome: Change From Baseline in CogState CPAL on Day 6
Description: as for outcome 7
Time Frame: Baseline and Day 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Errors
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Errors | 6.7933 (9.8653) | -16.7905 (9.8715) | 58.2002 (10.0337) | 3.1304 (9.9948)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7707, ANCOVA; LS Mean Difference = 3.6629, 95% CI 2-sided [-21.4729 to 28.7987], Standard Error of Mean 12.4945
Statistical Analysis 2: Comparison: Fesoterodine 8 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1162, ANCOVA; LS Mean Difference = -19.9210, 95% CI 2-sided [-44.9634 to 5.1215], Standard Error of Mean 12.4482

9. Secondary Outcome: CogState Groton Maze Learning Task (GMLT)
Description: GMLT: a cognitive test which assessed executive function. Participant was shown a 10 x 10 grid of tiles on a computer touch screen. A 28-step pathway was hidden among 100 possible locations. The participant was instructed to move 1 step from the start location and then continue 1 tile at a time, toward the end to find the pathway. The outcome measure was total number of errors made in attempting to learn the same hidden pathway on 5 consecutive trials at a single session. Lower scores meant a better performance.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Errors | 53.72 (17.091) | 58.39 (15.170) | 56.83 (15.023) | 52.28 (15.736)

10. Secondary Outcome: Change From Baseline in CogState Groton Maze Learning Task on Day 6
Description: as for outcome 9
Time Frame: Baseline and Day 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Errors
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Errors | -4.1399 (4.2079) | -5.7717 (4.2515) | 24.7115 (4.2033) | -4.1467 (4.2413)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9989, ANCOVA; LS Mean Difference = 0.0068, 95% CI 2-sided [-9.8297 to 9.8433], Standard Error of Mean 4.8707
Statistical Analysis 2: Comparison: Fesoterodine 8 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7485, ANCOVA; LS Mean Difference = -1.6251, 95% CI 2-sided [-11.7926 to 8.5425], Standard Error of Mean 5.0346

11. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: RAVLT evaluates a wide diversity of functions: short-term auditory-verbal memory, rate of learning, learning strategies, retroactive, and proactive interference, presence of confabulation of confusion in memory processes, retention of information, and differences between learning and retrieval. Assessment of RAVLT is between 10 to 15 minutes; Performance variable: the sum of the number of words recalled successfully on the delayed recall trial. Higher score meant a better performance.
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Words Recalled
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Words Recalled | 6.50 (3.884) | 6.67 (3.630) | 7.22 (3.687) | 6.33 (3.378)

12. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT) on Day 6
Description: as for outcome 11
Time Frame: Baseline and Day 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Words Recalled
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 18 | 18
Words Recalled | 0.1565 (0.5825) | -0.1780 (0.5820) | -3.9222 (0.5890) | -0.1119 (0.5862)
Statistical Analysis 1: Comparison: Fesoterodine 4 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7458, ANCOVA; LS Mean Difference = 0.2684, 95% CI 2-sided [-1.3788 to 1.9157], Standard Error of Mean 0.8243
Statistical Analysis 2: Comparison: Fesoterodine 8 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.9366, ANCOVA; LS Mean Difference = -0.0661, 95% CI 2-sided [-1.7202 to 1.5880], Standard Error of Mean 0.8277

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine 4 mg | Fesoterodine 8 mg | Aplrazolam 1 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 11/19 | 18/19 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 mg (N=20) | Fesoterodine 8 mg (N=19) | Aplrazolam 1 mg (N=19) | Placebo (N=20)
Dry eye (Eye disorders) | 0 | 1 | 1 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 6 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 4 | 1
Headache (Nervous system disorders) | 1 | 2 | 2 | 3
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 10 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.